CLINICAL TRIAL: NCT04223895
Title: Phase I Clinical Trial to Compare the Pharmacokinetics and Tolerability of CKD-386 With Co-administration of D012, D326, and D337 in Healthy Adult Volunteers
Brief Title: A Clinical Trial to Investigate the Pharmacokinetics and Safety/Tolerability of CKD-386 in Healthy Adult Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A83_04BE1917P
Record Dates: First submitted 2020-01-08; First posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Type2 Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1 (Experimental): Period 1: D012, D326, D337(3 tabs, once) / Period 2: CKD-386 F1(1 tab, once)/ Period 3: CKD-386 F2(1 tab, once)
  Interventions: Drug: CKD-386 Formulation 1; Drug: CKD-386 Formulation 2; Drug: D012, D326 and D337
- Group 2 (Experimental): Period 1: D012, D326, D337(3 tabs, once) / Period 2: CKD-386 F2(1 tab, once)/ Period 3: CKD-386 F1(1 tab, once)
  Interventions: Drug: CKD-386 Formulation 1; Drug: CKD-386 Formulation 2; Drug: D012, D326 and D337
- Group 3 (Experimental): Period 1: CKD-386 F1(1 tab, once) / Period 2: D012, D326, D337(3 tabs, once) Period 3: CKD-386 F2(1 tab, once)
  Interventions: Drug: CKD-386 Formulation 1; Drug: CKD-386 Formulation 2; Drug: D012, D326 and D337
- Group 4 (Experimental): Period 1: CKD-386 F1(1 tab, once) / Period 2: CKD-386 F2(1 tab, once) / Period 3: D012, D326, D337(3 tabs, once)
  Interventions: Drug: CKD-386 Formulation 1; Drug: CKD-386 Formulation 2; Drug: D012, D326 and D337
- Group 5 (Experimental): Period 1: CKD-386 F2(1 tab, once) / Period 2: D012, D326, D337(3 tabs, once)/ Period 3: CKD-386 F1(1 tab, once)
  Interventions: Drug: CKD-386 Formulation 1; Drug: CKD-386 Formulation 2; Drug: D012, D326 and D337
- Group 6 (Experimental): Period 1: CKD-386 F2(1 tab, once) / Period 2: CKD-386 F1(1 tab, once) / Period 3: D012, D326, D337(3 tabs, once)
  Interventions: Drug: CKD-386 Formulation 1; Drug: CKD-386 Formulation 2; Drug: D012, D326 and D337

INTERVENTIONS:
Drug: CKD-386 Formulation 1 — A single oral dose of 1 tablet under fasting conditions for each period
  Other Names: CKD-386 F1
Drug: CKD-386 Formulation 2 — A single oral dose of 1 tablet under fasting conditions for each period
  Other Names: CKD-386 F2
Drug: D012, D326 and D337 — A single oral dose of 3 tablets(D012, D326 and D337) under fasting conditions for each period

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and Safety/Tolerability of CKD-386

DETAILED DESCRIPTION:
Phase I clinical trial to compare the pharmacokinetics and tolerability of CKD-386 with co-administration of D012, D326, and D337 in healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Those who are over 19 years old at the screening visit
2. Those who weigh more than 50kg (45kg or more for women) at the screening visit and have a body mass index (BMI) within the range of 18-30kg/m^2
3. Those who meet the following conditions of blood pressure measured in a sitting position after sufficient rest at the screening visit

   * Systolic blood pressure: 90mmHg or more and 139mmHg or less
   * Diastolic blood pressure: 60mmHg or more and 89mmHg or less
4. Those who no congenital or chronic disease based on screening and no pathological symptoms or findings in medical examination results (e.g. EEG, ECG, chest and gastroscopy or gastrointestinal radiographs, if necessary)
5. The person in charge of the examination (or authorized test physician) who has determined that the test subject is suitable for the diagnostic test and electrocardiogram test such as hematology test, blood chemistry test, serology test and urine test performed according to the characteristics of the investigational drug product
6. Persons agreeing to exclude the possibility of pregnancy using appropriate contraceptive methods and not providing sperm or eggs from the date of first administration of the investigational drug to the 14th day after the last administration of the investigational drug

Exclusion Criteria:

1. Those who participated in other clinical trials (including bioequivalence studies) within 6 months before the first dose and received the investigational drug
2. Those who used drugs that induce and inhibit metabolic enzymes, such as barbital drugs, within one month before the first dose, or who used drugs that may interfere with this test within 10 days before the first dose
3. Those who have donated whole blood within 2 months before the first dose or component donation within 1 month, or have transfused within 1 month
4. Those who have had a history of gastrointestinal resection that may affect the absorption of the investigational drug (except appendectomy and hernia surgery)
5. A person who meets the following conditions within one month before the first administration date

   * Excess alcohol: 21 cups / week for men and 14 cups / week for women.

     [1 glass = 50 mL of shochu or 30 mL of liquor or 250 mL of beer]
   * Smokers exceeding 20 cigarettes per day
6. Patients with the following diseases

   * Patients with hypersensitivity to the main constituents or components of the investigational drug
   * Severe hepatic impairment, biliary atresia or cholestasis
   * Patients with hereditary angioedema or with a history of angioedema in the treatment of ACE inhibitors or angiotensin II receptor antagonists
   * Diabetes mellitus
   * Patients with moderate to severe renal impairment [glomerular filtration rate (eGFR) <60 mL / min / 1.73m^2]
   * Renal vascular hypertension patients
   * Patients with active liver disease, including unexplained persistent serum transaminase elevations or elevated serum transaminase elevations greater than three times the normal upper limit
   * Patients with myopathy or have a history of family or genetic history of myopathy
   * Hypothyroidism
   * If you have a history of muscle toxicity for other HMG-CoA converting enzymes or fibrate class drugs
7. Genetic problems such as galactose intolerance, Lapp lactose deficiency, or glucose-galactose malabsorption
8. person who is considered to be unsuitable for participation in this clinical trial for reasons other than the above selection / exclusion criteria.
9. In the case of female volunteers, the suspected or lactating woman

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-03-04 (Estimated); Study Completion 2020-06-15 (Estimated)

PRIMARY OUTCOMES:
AUCt of each main component or metabolite of the component after single dose of CKD-386 F1, CKD-386 F2 and D012, D326, D337 | 0(predose)~72 hours
  AUCt: Area under the concentration-time curve
Cmax of each main component or metabolite of the component after single dose of CKD-386 F1, CKD-386 F2 and D012, D326, D337 | 0(predose)~72 hours
  Cmax: Maximum plasma concentration of the drug

SECONDARY OUTCOMES:
AUCinf each main component or the metabolite of the component after single dose of CKD-386 F1, CKD-386 F2 and D012, D326, D337 | 0(predose)~72 hours
  AUCinf: Area under the concentration-time curve from zero up to ∞
tmax each main component or the metabolite of the component after single dose of CKD-386 F1, CKD-386 F2 and D012, D326, D337 | 0(predose)~72 hours
  tmax: Time to maximum plasma concentration
AUCt/AUCinf each main component or the metabolite of the component after single dose of CKD-386 F1, CKD-386 F2 and D012, D326, D337 | 0(predose)~72 hours
  AUCt/AUCinf: AUCt/AUCinf Ratio
t1/2 each main component or the metabolite of the component after single dose of CKD-386 F1, CKD-386 F2 and D012, D326, D337 | 0(predose)~72 hours
  t1/2: Terminal elimination half-life
AUCt of each main component or metabolite of the component after single dose of CKD-386 F1, CKD-386 F2 and D326, D337 | 0(predose)~72 hours
  AUCt: Area under the concentration-time curve
Cmax of each main component or metabolite of the component after single dose of CKD-386 F1, CKD-386 F2 and D326, D337 | 0(predose)~72 hours
  Cmax: Maximum plasma concentration of the drug

CONTACTS AND LOCATIONS:
Overall Officials: 70-4665-9174 70-4665-9174, Principal Investigator — H Plus Yangji Hospital